CLINICAL TRIAL: NCT04566718
Title: A Treatment Legacy Effect of Metformin on Metabolic and Endocrine Parameters in Obese Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: A Treatment Legacy Effect of Metformin in Obese Women With PCOS
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, Clinical Professor, University Medical Centre Ljubljana
Other Study IDs: MET prosp
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: PCOS
Keywords: PCOS; obesity; metformin
MeSH Terms: conditions — Obesity | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Obese women who have been treated with metformin for one year prior to the study.
  Interventions: Drug: Metformin
- Group B: Obese women who have been treated with metformin for at least three years prior to the study.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — metformin cessation

SUMMARY:
Metformin has multiple health promoting effects and it may serve as a preventive measure for individuals who are at high risk for metabolic complications.

According to the latest international guidelines it should be considered as an adjunct therapy to lifestyle intervention in all overweight/obese women with PCOS, independently of their glucose homeostasis and menstrual regularity. However, there is no clear answer for how long metformin should be prescribed in this subset of women with PCOS and for how long the beneficial impact would sustain after treatment cessation.

The investigators compared the consequences of metformin withdrawal after long-term therapy as opposed to the consequences of metformin suspension after short term therapy in overweight/obese women with PCOS that had previously responded to metformin by means of moderate weight loss, improved menstrual frequency and sustained normal glucose homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* PCOS defined by the National Institute of Child Health and Human Development (NICHD) criteria
* obesity with body mass index ≥ 30 kg/m2
* normal glucose homeostasis at metformin treatment

Exclusion Criteria:

* known type 1 or type 2 diabetes mellitus
* heart failure
* renal insufficiency with serum creatinine more than 125 umol/L
* arterial hypertension
* pregnancy
* BMI below 25 kg/m2

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: The investigators conducted 20 obese women with PCOS with normal glucose homeostasis (without known type 1 or type 2 diabetes mellitus) who have been treated with metformin for one year prior to the study and 20 obese women with PCOS with normal glucose homeostasis (without known type 1 or type 2 diabetes mellitus) who have been treated with metformin for at least three years prior to the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
The main outcome was change in body weight. | Patient's body weight was measured at the base point and at the endpoint of 6 months of clinical trial.
The main outcome was change in insulin resistance measured with homeostasis model assessment (HOMA IR). | HOMA IR was calculated at the base point and at the endpoint of 6 months of clinical trial.
  HOMA IR was calculated as the product of the fasting glucose and insulin concentration divided by 22.5.
The main outcome was change in expression of glucose transporter type 4 (GLUT-4) in adipose tissue. | We did adipose tissue needle biopsy at the base point and at the endpoint of 6 months of clinical trial. All samples were frozen and then analysed together after end point of the study.
  We obtained adipose tissue using needle biopsy, from which we isolated ribonucleic acid and after reverse transcription, real-time quantitative polymerase chain reaction determined messenger ribonucleic acid expression for GLUT-4.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Kravos NA, Janez A, Goricar K, Dolzan V, Jensterle M. Effects of metformin withdrawal after long and short term treatment in PCOS: observational longitudinal study. Diabetol Metab Syndr. 2021 Apr 12;13(1):43. doi: 10.1186/s13098-021-00660-5. PMID 33845893